CLINICAL TRIAL: NCT05247294
Title: Assessment of Fluctuating Parkinson's Disease With Sensor-based Home Monitoring
Status: Completed | Type: Observational
Sponsor: Sheba Medical Center (Other Government)
Collaborators: AbbVie (Industry); Intel Electronics Ltd. (Unknown)
Responsible Party: Principal Investigator, Dr. Sharon Hassin, Prof. Sharon Hassin, Sheba Medical Center
Other Study IDs: 5428-18
Record Dates: First submitted 2022-01-26; First posted 2022-02-18 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease; Home based monitoring; Sensor-based data; Motor fluctuations
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to implement home-based monitoring (HBM) using remote-capture wearable devices and patient reported outcomes (PROs) in a rather homogeneous subgroup of advanced Parkinson's Disease (PD) patients, suffering from significant motor fluctuations (MF) and Levodopa-induced dyskinesia (LID), over a two-week period.

The investigators aim to provide a more comprehensive picture of patient symptoms, severity, and fluctuations and compare these data to interview-derived clinical data.

DETAILED DESCRIPTION:
Parkinson's Disease (PD) is a neuro-degenerative disorder affecting millions of people worldwide. PD is associated with both motor and non-motor symptoms that affect patients' functioning and Quality of life.

The motor symptoms consist of tremor, rigidity, bradykinesia and gait impairments. Additional important motor symptoms that are associated with chronic Levodopa therapy, are levodopa-induced dyskinesia and motor fluctuations.

Currently, the accepted clinical measurement of PD symptom severity is the Movement Disorders Society-unified Parkinson's disease rating scale (MDS-UPDRS), which is based, in part, on subjective and potentially recall-based reports by the patients and on semi-objective observations by the clinician.

On average, PD patients see their treating neurologist for in-clinic visits twice a year. These visits are limited in time and may leave some issues unattended regarding all aspects of disease and overall health. This may adversely affect the decision making process and the prescribed treatment plan.

In order to understand the accurate clinical status of patients, particularly in the motor fluctuating stage of PD and to monitor results of intervention, the treating neurologist may need a more comprehensive picture of their patients' symptoms and lives during protracted periods and real life in their home environment.

The HBM apparatus used in this study will consist of a smartwatch (Apple watch) and a smartphone (Apple iPhone 8). The phone is pre-installed with an application which is part of the Intel® Pharma Analytics Platform. The mobile app was designed by usability experts and was tested with patients to ensure ease of use by an elderly population with PD.

The Intel platform is enhanced by a compendium of algorithms to extract clinical insights from the raw sensor data. Passive sensor data is transferred from the study smartwatch. The data includes three measures based on the smartwatch data: activity level, dyskinesia and tremor.

The study will be conducted at Movement Disorders Institute at Sheba Medical Center and will include two clinic visits and a 2-week HBM phase.

The first clinic visit as well as the 2-week home period will include the following daily assessments (once in "off" state and once in "on" state):

1. 3- meter Timed up and go test (3mTUG)
2. Finger tapping on smartphone (10 seconds, both hands)
3. Hand tremor assessment: postural tremor (outstretched, 30 sec), rest tremor (30 sec)
4. Pronation-supination

In addition, ePROs are captured with electronic home diaries. Participants will report the severity of PD symptoms they are experiencing on a 5-point scale throughout the day. For the duration of waking hours, participants will receive a notification on their phone to input information about their ON/OFF state every 30 minutes.

The primary objective is to correlate severity of fluctuating motor symptoms in PD patients using the Intel® Pharma Analytics Platform's derived passive sensor data (percentage of daily tremor time and percentage of daily dyskinesia time, percentage of daily "inactivity") in an exploratory manner with concomitant assessment of motor fluctuations and dyskinesia using the application's based electronic symptom diary and data of tremor, off time and dyskinesia using the MDS-UPDRS scale.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of idiopathic Parkinson's disease for at least 5 years
2. Males or females over the age of 30
3. Patients treated with oral levodopa (3 daily doses or more), reporting motor fluctuations and (preferably) with l-dopa-induced dyskinesia
4. UPDRS-MDS 4.4 functional impact of fluctuations (mild + severe, 2-4)
5. Hoehn &Yahr stage 1-3 while ON
6. Ability to operate smartphone technology in the household
7. Mini-Mental State Examination score >20

Exclusion Criteria:

1. Cognitive or psychiatric impairment that would preclude study participation as determined by the principal investigator
2. Additional major comorbidities
3. Levodopa-resistant tremor (tremor during ON)
4. Levodopa-resistant freezing (freezing during ON)
5. Previous surgical treatment for PD

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Advanced Parkinson's Disease (PD) patients, suffering from significant motor fluctuations (MF) and Levodopa-induced dyskinesia (LID)
Sampling Method: Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2019-11-03 (Actual); Primary Completion 2021-02-24 (Actual); Study Completion 2021-02-24 (Actual)

PRIMARY OUTCOMES:
Correlation between sensor data and MDS-UPDRS data | 2-3 weeks study period
  To correlate severity of fluctuating motor symptoms in PD patients using Intel® Pharma Analytics Platform's derived passive sensor data (percentage of daily tremor time and percentage of daily dyskinesia time, percentage of daily "inactivity") in an exploratory manner with concomitant assessment of motor fluctuations and dyskinesia using the application's based electronic symptom diary and data of tremor, off time and dyskinesia using the MDS-UPDRS.

SECONDARY OUTCOMES:
Correlation between passive sensor data and PDQ-39 questionnaire | 2-3 weeks study period
  Correlate the results of passive sensor data regarding "level of activity" and "time of activity" with measures of Quality of life as captured by the PDQ-39
Correlation between passive sensor data and electronic home diaries | 2-3 weeks study period
  Correlate the results passive sensor data of "level of activity" and "time of activity" with "on" and "off" data obtained from electronic home diary (on the same days).
Correlation between motor test results (TUG, Static postural tests and finger tapping,) and relevant MDS-UPDRS items | 2-3 weeks study period
  Correlate the results of guided structured motor tests (TUG, Static postural tests and finger tapping,) during "off" and during "on" performed in the clinic (visit 1) and at home (twice in each condition) with the results of in-clinic MDS-UPDRS items: 3.1 walking, 3.11 freezing of gait, 3.12 postural stability, 3.4 finger taps during "off" and during "on"
Assessing compliance of PD patients using wearable devices and adherence to assessment protocol. | 2-3 weeks study period
  The measures consist of: overall use of watch, Diary report -delay, Number of skipped daily questionnaires, number of skipped assessments, number of skipped medication reports, number of delayed medication reports, number of skipped medications intake, delay in medication intake and more.
Correlation between medication regimen as prescribed by neurologist and patient adherence in real life | 2-3 weeks study period
  To correlate medication regimen as prescribed by neurologist and patient adherence in real life, using electronic medication intake reporting

CONTACTS AND LOCATIONS:
Locations (1):
- Movement Disorders Institution, Sheba Medical Center, Ramat Gan, Israel